CLINICAL TRIAL: NCT02687555
Title: The Role of Computerized Training in Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Daimler und Benz Stiftung (Unknown); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Marcella Woud, Postdoctoral Research Fellow, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32-12/14; 204 (Other: Fakultät für Psychologie Ethikkommission, Ruhr University of Bochum); 15-5477 (Other: Ethik-Kommission der Medizinischen Fakultät, Ruhr University of Bochum)
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Computerized Cognitive Bias Modification of Appraisals (CBM-App), developed from that used by Woud et al. (2012,2013). The intervention comprises 8 sessions completed over a period of 2 weeks. The training takes place while participants are also receiving specialized inpatient treatment for PTSD at the Clinic for Psychosomatic Medicine and Psychotherapy, LWL University Clinic of Ruhr University of Bochum.
  Interventions: Behavioral: Cognitive Bias Modification of Appraisals (CBM-App)
- Control (Sham Comparator): Computerized Peripheral Vision Task (PVT), developed from that used by Calkins et al. (2015). The intervention comprises 8 sessions completed over a period of 2 weeks. The training takes place while participants are also receiving specialized inpatient treatment for PTSD at the Clinic for Psychosomatic Medicine and Psychotherapy, LWL University Clinic of Ruhr University of Bochum.
  Interventions: Behavioral: Peripheral Vision Task (control condition)

INTERVENTIONS:
Behavioral: Cognitive Bias Modification of Appraisals (CBM-App)
  Arms: Intervention
Behavioral: Peripheral Vision Task (control condition)
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether a computerized training, "Cognitive Bias Modification" targetting appraisals (CBM-App), can reduce dysfunctional appraisals of trauma in patients with Post-Traumatic Stress Disorder (PTSD), compared to a control condition. Other outcomes measured include symptoms of PTSD and trauma-relevant dysfunctional cognitions. Participants are recruited from inpatients with PTSD admitted to the Clinic for Psychosomatic Medicine and Psychotherapy, LWL University Clinic of Ruhr University of Bochum.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Post-Traumatic Stress Disorder according to ICD-10 (F43.1), and DSM-5 (as assessed via Clinician Adminstered PTSD Scale for DSM-5)
* motivated and willing to take part in the study (including questionnaire measures, computer training, filling out questionnaires after discharge)
* aged 18-60 years, male or female
* fluent in German

Exclusion Criteria:

* Substance abuse/ substance dependence currently or in the past six months
* active suicidal thoughts or intentions
* psychotic disorder (past or present)
* learning disability/ intellectual impairment
* red-green colour blindness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Dysfunctional trauma-related appraisals as measured using an open-ended ambiguous scenarios task | Post-intervention (~ 2 weeks post-baseline)

SECONDARY OUTCOMES:
Dysfunctional trauma-related appraisals as measured using an open-ended ambiguous scenarios task | Baseline, Mid-intervention (~1 week post-baseline), End of inpatient admission (~6 weeks post-baseline), 6 weeks post-discharge, 3 months post-discharge
Post-Traumatic Cognitions Inventory (PTCI) | Baseline, Mid-intervention (~1 week post-baseline), Post-intervention (~2 weeks post-baseline), End of inpatient admission (~6 weeks post-baseline), 6 weeks post-discharge, 3 months post-discharge
  The PTCI (Foa et al., 1999) is administered asking participants to report on their experience of post-traumatic cognitions in the previous week.
PTSD Checklist for DSM-5 (PCL-5) | Baseline, Mid-intervention (~1 week post-baseline), Post-intervention (~2 weeks post-baseline), End of inpatient admission (~6 weeks post-baseline), 6 weeks post-discharge, 3 months post-discharge
  The PCL-5 (Weathers et al., 2013; German version by Ehring, Knaevelsrud, Krüger & Schäfer) is administered asking participants to report on their experience of post-traumatic symptoms in the previous week.
Intrusions Questionnaire | Baseline, Mid-intervention (~1 week post-baseline), Post-intervention (~2 weeks post-baseline), End of inpatient admission (~6 weeks post-baseline), 6 weeks post-discharge, 3 months post-discharge
  The intrusions questionnaire asks participants to report on the frequency and characteristics of intrusive memories of trauma in the preceding week
Trauma Implicit Associations Test (IAT) | Baseline, Post-intervention (~2 weeks post-baseline)
  As developed by Lindgren et al. (2013)

OTHER OUTCOMES:
Hair Cortisol Concentration | Baseline, End of inpatient admission (~6 weeks post-baseline), 3 months post-discharge
Participant Feedback Questionnaire | 3 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcella L Woud, PhD, Principal Investigator — Ruhr University of Bochum
Locations (1):
- Clinic for Psychosomatic Medicine and Psychotherapy, LWL University Clinic of Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make individual participant data available on publication of the associated study results, via a publically-available data repository such as Open Science Framework. Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.

REFERENCES:
- [Derived] Woud ML, Blackwell SE, Cwik JC, Margraf J, Holmes EA, Steudte-Schmiedgen S, Herpertz S, Kessler H. Augmenting inpatient treatment for post-traumatic stress disorder with a computerised cognitive bias modification procedure targeting appraisals (CBM-App): protocol for a randomised controlled trial. BMJ Open. 2018 Jun 30;8(6):e019964. doi: 10.1136/bmjopen-2017-019964. PMID 29961004